CLINICAL TRIAL: NCT03777397
Title: Study of Awareness of Hospices Civils de Lyon Workers About Breast Cancer Screening
Brief Title: Awareness About Breast Cancer Screening
Acronym: DEPSEIN_HCL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0769
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire on the level of awareness of this risk among health sector employees, and more specifically the Lyon Civilian Hospices, and on participation in breast cancer screening for HCL employees, particularly among night shift staff.

SUMMARY:
Breast cancer is the most common cancer in French women, with 52000 new cases each year.

Shift work and night work is recognized by International Agency for Research on Cancer as a potential risk factor. Epidemiological studies find, for most of them, an increased risk of breast cancer compared with general population. Physiological hypothesis rely on the melatonin role in defense against tumorigenesis.

According to High Authority of Health clinical good practice guidelines, the risk does not justify more screening than the organized screening. We do not have information about awareness level of workers in health structures, specially in the Hospices Civils de Lyon.

Investigators would like to know how employees take part to breast cancer screening, specially in night workers.

This study, as a survey, is a first step to evaluate the need for specific actions to increase the participation to breast cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* employees HCL
* women

Exclusion Criteria:

* <18 years old

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women employees of Hospices Civils de Lyon
Sampling Method: Non-Probability Sample
Enrollment: 2264 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Participation of HCL female staff in mammography screening for breast cancer | 5 minutes
  One question of the questionnaire is about this participation

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie - Hôpital de la Croix-Rousse - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No